CLINICAL TRIAL: NCT03510650
Title: Diagnostic Biomarkers for Adult Hemophagocytic Lymphohistiocytosis in Critically Ill Patients (HEMICU)
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Operative Intensive Care Medicine (CCM, CVK), Charité - Universitätsmedizin Berlin, Charite University, Berlin, Germany
Other Study IDs: HEMICU
Record Dates: First submitted 2018-04-05; First posted 2018-04-27 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Hemophagocytic Lymphohistiocytosis
Keywords: Hemophagocytic Lymphohistiocytosis (HLH); Hemophagocytic syndrome (HPS); critically ill; Intensive care unit (ICU)
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 6 ml of blood samples of each patient will be stored in the Biobank of the Berlin Institute of Health, Clinical Research Unit, Charité - Universitätsmedizin Berlin, Campus Virchow-Klinikum, Augustenburger Platz 1, D-13353 Berlin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: 50 patients with sepsis versus 50 patients with HLH [anticipated]

SUMMARY:
Hemophagocytic lymphohistiocytosis in adults (HLH) is at 68% mortality whereas 78% of all cases remain undiagnosed though therapies are available which clearly reduce mortality. The investigators aim to systematically investigate this life-threatening hyperinflammatory syndrome in intensive care units (ICU) in order to detect biomarkers that are highly sensitive and highly specific for HLH in ICU compared to patients with sepsis.

DETAILED DESCRIPTION:
The investigators will draw blood samples of 100 patients at the time of diagnosis (each 50 with suspected or diagnosed HLH/sepsis) to determine a cytokine panel (c reactive protein (CRP), procalcitonin (PCT), interleukin (IL) 1β, IL-6, IL-8, IL-10, IL-18, IL-33, tumor necrosis factor (TNF) α, interferon (IFN) ɣ, soluble IL-2 receptor (sIL-2R), the EBV and CMV viral loads, human immunodeficiency virus (HIV) antibodies and -antigen, perforin, fibrinogen, triglycerides, bilirubin, lactate dehydrogenase, liver transaminases, sodium, serum albumin, electrophoresis, glycosylated ferritin, the microRNAs miR-205-5p, miR-194-5p and miR-30c-5p, perforin, CD107a and high immune status (differential blood count, T cells, B cells, NK cells, T helper cells, cytotoxic T cells, CD4 / CD8 ratio, HLA-DR of CD8 +, CD11a of CD8, CD57 of CD8, CD28 of CD8 +, HLA-DR of monocytes, CD56bright and CD69 of NK cells). The results of this study serve the development of new clinical concepts in order to safely diagnose HLH at an early stage, to distinguish from sepsis and to reduce the fatal consequences.

ELIGIBILITY:
Inclusion Criteria:

* Male or female critically ill patients
* At least 18 years old
* Suspected or diagnosed HLH

Exclusion Criteria:

* Female patients: Pregnancy
* Female patients: Breastfeeding

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female critically ill patients admitted to any ICU of the Charité - Universitätsmedizin Berlin.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2022-06-26 (Actual); Study Completion 2022-12-26 (Actual)

PRIMARY OUTCOMES:
Incidence of HLH in intensive care units based on HLH-2004 criteria | Up to 180 days
  HLH patients are followed up until the end of hospital stay or death.

SECONDARY OUTCOMES:
Intensive care unit stay | Participants will be followed up for the duration of hospital length of stay, an expected average of 4 weeks
Hospital stay | Participants will be followed up for the duration of hospital length of stay, an expected average of 8 weeks
Mortality | Up to 180 days
  Mortality after 30 and 180 days
Cytokine panel | Up to 180 days
  1 blood sample of Cytokine panel (CRP, PCT, IL-1β, IL-6, IL-8, IL-10, IL-18, IL-33, TNF-α, IFN-ɣ, sIL-2R, ferritin) collection at time of diagnosed HLH
Epstein Barr Virus (EBV) and Cytomegalovirus (CMV) viral loads | Up to 180 days
  1 blood sample collection at time of diagnosed HLH
Glycosylated ferritin | Up to 180 days
  1 blood sample collection at time of diagnosed HLH
microRNAs miR-205-5p, miR-194-5p and miR-30c-5p | Up to 180 days
  1 blood sample collection at time of diagnosed HLH
Perforin and CD107a | Up to 180 days
  1 blood sample collection at time of diagnosed HLH
Human immunodeficiency virus antibodies and -antigen | Up to 180 days
  1 blood sample collection at time of diagnosed HLH
Fibrinogen | Up to 180 days
Triglycerides | Up to 180 days
Bilirubin | Up to 180 days
Lactate dehydrogenase | Up to 180 days
  Lactate dehydrogenase is measured in U/l
Liver transaminase (ASAT) | Up to 180 days
  ASAT [U/l]
Liver transaminases (ALAT) | Up to 180 days
  ALAT [U/l]
Sodium | Up to 180 days
Serum albumin | Up to 180 days
Serum protein electrophoresis | Up to 180 days
  Serum protein Electrophoresis (%) is used to separate and quantify the serum protein components into serum albumin, alpha-1 globulins, alpha-2 globulins, beta 1 and 2 globulins, and gamma Globulins.
Detailed immune status | Up to 180 days
  The immune status is analyzed by differential blood count [/nl], T cells [/nl], B cells [/nl], NK cells [/nl], T helper cells [/nl], cytotoxic T cells [/nl], CD4 / CD8 ratio, HLA-DR of CD8+ [%], CD11a of CD8 [%], CD57 of CD8 [%], CD28 of CD8+ [%], HLA-DR of monocytes [antigen/cell], CD56bright [%] and CD69 [%] of NK cells.

OTHER OUTCOMES:
HLA Typing | At the beginning of the investigation
  HLA testing identifies the major HLA genes a person has inherited and their corresponding antigens that are present on the surface of their cells.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicine (CCM, CVK), Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barba T, Maucort-Boulch D, Iwaz J, Bohe J, Ninet J, Hot A, Lega JC, Guerin C, Argaud L, Broussolle C, Jamilloux Y, Richard JC, Seve P. Hemophagocytic Lymphohistiocytosis in Intensive Care Unit: A 71-Case Strobe-Compliant Retrospective Study. Medicine (Baltimore). 2015 Dec;94(51):e2318. doi: 10.1097/MD.0000000000002318. PMID 26705219
- [Derived] Lachmann G, Knaak C, von Haefen C, Paeschke N, Meisel C, Nyvlt P, Schuster FS, Piper SK, Kruppa J, Vorderwulbecke G, Balzer F, La Rosee P, Schenk T, Unterwalder N, Kolsch U, Lachmann N, Akyuz L, Brunkhorst FM, Volk HD, Keh D, Spies C. Diagnostic biomarkers for adult haemophagocytic lymphohistiocytosis in critically ill patients (HEMICU): a prospective observational study protocol. BMJ Open. 2019 Oct 30;9(10):e032695. doi: 10.1136/bmjopen-2019-032695. PMID 31666276